CLINICAL TRIAL: NCT00413023
Title: A Randomised, Double-Blind, Double-Dummy, Parallel-Group, Placebo-Controlled, Forced Dose Titration Study Evaluating the Efficacy and Safety of GW679769 and Paroxetine in Subjects With Major Depressive Disorder (MDD)
Brief Title: Study Of The Effects Of A New Antidepressant Therapy In Patients With Major Depressive Disorder (MDD)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NKF100096
Record Dates: First submitted 2005-08-24; First posted 2006-12-19 (Estimated); Last update posted 2016-10-28 (Estimated); Status verified 2016-10

CONDITIONS: Depressive Disorder, Major
Keywords: depression; major depressive disorder; MDD
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — casopitant

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: GW679769

SUMMARY:
The purpose of this study is to assess the efficacy, safety and tolerability of GW679769 patients with Major depressive Disorder (MDD).

ELIGIBILITY:
Inclusion criteria:

* Primary diagnosis of Major depressive Disorder as defined in DSM-IV.
* Capable of giving informed consent and willing to comply with the study requirements.
* Women of childbearing potential must agree to one of a number of defined acceptable methods of birth control.

Exclusion Criteria:

* Primary diagnosis within the past 6 months of another Axis 1 disorder such as an anxiety disorder.
* Use of medications for a psychiatric condition including herbals in the past 2-12 weeks according to medication type.
* Subjects who, in the investigator's judgement, pose a current, serious suicidal or homicidal risk or have made a suicide attempt within the past 6 months.
* Subjects who currently meet or who met within 6 months prior to screening DSM-IV criteria for substance abuse or subjects who currently meet or who met within 6 months prior to screening DSM-IV criteria for substance dependence (other than nicotine).
* Significantly abnormal blood or urine laboratory tests or electrocardiogram (ECG).

Ages: 18 Years to 64 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 348 (Actual)
Dates: Start 2005-06; Primary Completion 2006-09 (Actual); Study Completion 2006-09 (Actual)

PRIMARY OUTCOMES:
Change in score on a Depression rating scale following 8 weeks of treatment.

SECONDARY OUTCOMES:
Change in score on a number of rating scales following 8 weeks of treatment assessing symptomatic, behavioural and functional parameters which together provide a more complete description of the disorder.

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (34):
- Argentina (3):
  - GSK Investigational Site, Buenos Aires, Buenos Aires
  - GSK Investigational Site, Córdoba, Córdoba Province
  - GSK Investigational Site, Buenos Aires
- Belgium (4):
  - GSK Investigational Site, Alken
  - GSK Investigational Site, Kortrijk
  - GSK Investigational Site, Liège
  - GSK Investigational Site, Mont-Godinne
- Chile (2):
  - GSK Investigational Site, Providencia / Santiago, Región Metro de Santiago
  - GSK Investigational Site, Santiago, Región Metro de Santiago
- Costa Rica (2):
  - GSK Investigational Site, San José, Provincia de San José
  - GSK Investigational Site, San José
- Germany (8):
  - GSK Investigational Site, Ellwangen, Baden-Wurttemberg
  - GSK Investigational Site, Würzburg, Bavaria
  - GSK Investigational Site, Hüttenberg, Hesse
  - GSK Investigational Site, Achim, Lower Saxony
  - GSK Investigational Site, Bochum, North Rhine-Westphalia
  - GSK Investigational Site, Hattingen, North Rhine-Westphalia
  - GSK Investigational Site, Dresden, Saxony
  - GSK Investigational Site, Berlin, State of Berlin
- Italy (4):
  - GSK Investigational Site, Guardiagrele (CH), Abruzzo
  - GSK Investigational Site, Bologna, Emilia-Romagna
  - GSK Investigational Site, Milan, Lombardy
  - GSK Investigational Site, Pisa, Tuscany
- GSK Investigational Site, Lima, Peru
- Poland (3):
  - GSK Investigational Site, Bialystok
  - GSK Investigational Site, Chełmno
  - GSK Investigational Site, Kościan
- Slovakia (5):
  - GSK Investigational Site, Bratislava
  - GSK Investigational Site, Levoča
  - GSK Investigational Site, Liptovský Mikuláš
  - GSK Investigational Site, Rimavská Sobota
  - GSK Investigational Site, Trenčín
- GSK Investigational Site, Oviedo, Spain
- GSK Investigational Site, Solna, Sweden

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Ratti E, Bellew K, Bettica P, Bryson H, Zamuner S, Archer G, Squassante L, Bye A, Trist D, Krishnan KR, Fernandes S. Results from 2 randomized, double-blind, placebo-controlled studies of the novel NK1 receptor antagonist casopitant in patients with major depressive disorder. J Clin Psychopharmacol. 2011 Dec;31(6):727-33. doi: 10.1097/JCP.0b013e31823608ca. PMID 22020354
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: NKF100096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: NKF100096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: NKF100096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: NKF100096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: NKF100096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: NKF100096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: NKF100096 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register